CLINICAL TRIAL: NCT05706441
Title: Lung and Diaphragm Ultrasound Evaluation During Weaning From Mechanical Ventilation in COVID-19 Patients：A Prospective, Observational Study
Brief Title: Lung and Diaphragm Ultrasound Evaluation During Weaning From Mechanical Ventilation in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0017
Record Dates: First submitted 2023-01-18; First posted 2023-01-31 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-01

CONDITIONS: Weaning; COVID-19; Lung Ultrasound; Diaphragm Ultrasound
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ultrasound: Pulmonary and diaphragm ultrasound was evaluated within one hour before withdrawal
  Interventions: Other: Point-of-Care Ultrasound

INTERVENTIONS:
Other: Point-of-Care Ultrasound — Ultrasonographic scans of the lung and right hemidiaphragm were acquired after 30 min from the beginning of the SBT, or immediately before reconnecting the patient to the ventilator in the case of SBT failure occurring before

SUMMARY:
The goal of this observational study is to learn about the function of lung and diaphragm ultrasound during weaning from mechanical ventilation in COVID-19 patients. The aim of this study was that the lung ultrasound score and diaphragm muscle mobility could be a potential predictive factor of weaning success.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* critically ill patients with COVID-19 (defined as those requiring mechanical ventilation due to respiratory failure), and eligible for their first SBT according to the attending physician's judgement that the underlying disease which led to intubation had sufficiently resolved.

Exclusion Criteria:

* patients with previous cardiothoracic surgery or pleurodesis and patients who presented with stridor (due to upper airway involvement) as a cause of extubation failure
* neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: admission to a COVID-19 ICU with hypoxemic respiratory failure； start of weaning from mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
The primary end-point was to verify the lung and diaphragm ultrasound evaluation if the predicts weaning success/failure from mechanical ventilation | spontaneous-breathing trial started until 48 hours following extubation
  Weaning failure was defined as failure to pass the spontaneous-breathing trial or the need for re-intubation within 48 h following extubation

SECONDARY OUTCOMES:
The secondary outcome was to verify the predictive value of the traditional weaning parameters | spontaneous-breathing trial started until 48 hours following extubation
  Weaning failure was defined as failure to pass the spontaneous-breathing trial or the need for re-intubation within 48 h following extubation

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Yi Y, Zhang F, Yao YY, Chen YX, Wu CM, Wang RY, Yan M. Lung Ultrasound Score as a Predictor of Failure to Wean COVID-19 Elderly Patients off Mechanical Ventilation: A Prospective Observational Study. Clin Interv Aging. 2024 Feb 19;19:313-322. doi: 10.2147/CIA.S438714. eCollection 2024. PMID 38404479